CLINICAL TRIAL: NCT00279851
Title: Prevalence of Hypoglycemia and/or Hyperinsulinism/Hyperammonemia Syndrome in Patients With Idiopathic Seizures.
Brief Title: Blood Sugars in Children With Idiopathic Seizures.
Status: Withdrawn | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Other Study IDs: 05046
Record Dates: First submitted 2006-01-18; First posted 2006-01-20 (Estimated); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Seizures; Hypoglycemia; Hyperammonemia
Keywords: idiopathic seizure; hypoglycemia; hyperammonemia/hyperinsulinism syndrome
MeSH Terms: conditions — Seizures; Hypoglycemia; Hyperammonemia; Hyperinsulinemic hypoglycemia, familial, 6

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to determine if there is a significant percentage of children with the diagnosis of idiopathic seizures who have undiagnosed or unrecognized hypoglycemia (low blood sugar).

DETAILED DESCRIPTION:
Convulsive disorders are among the most frequently occurring neurologic conditions in children. Idiopathic seizures are the most common (67.6%) type of seizure seen in the 0-15 year age group. The highest incidence is in the first year of life. In the United States, 5 percent of individuals experience a seizure of some type by the age of 20.

Seizures have multiple etiologies. These include hypoglycemia, congenital causes, toxic/metabolic causes, infection, neoplasm, perinatal causes, and trauma. The medical evaluation often includes blood work, imaging of the brain, and performing an electroencephalogram. Currently, there is no consensus as to the work-up of children presenting with unprovoked seizures.

Hypoglycemia presents with a wide spectrum of symptoms and severity. In children, hypoglycemia can lead to seizures and coma. In neonates and infants, however, the symptoms are even more varied and nonspecific. They can include cyanotic spells, apnea, respiratory distress, refusal to feed, and myoclonic jerks. The varied symptoms of hypoglycemia make the disorder difficult to diagnose.

The study will have parents checking blood sugars for 14 days and a one time ammonia level. Blood sugar checks will be first thing in the morning and one hour after a meal. If the study identifies a subset of patients with idiopathic seizures who have hypoglycemia, this finding may have implications for future glucose screening recommendations.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria will be patients with idiopathic seizure disorders.
* The age range will be from birth to 17 years of age.
* Study subjects may be on anti-convulsants; the study does not alter current drug therapy.

Exclusion Criteria:

* The exclusion criteria includes patients with known causes of seizure disorders, including those with an underlying risk factor predisposing them to seizures. The risk factors are:

  1. congenital causes (CNS malformation, cerebral palsy)
  2. CNS infection toxic/known metabolic abnormality
  3. CNS neoplasm perinatal insults (birth trauma, asphyxia/hypoxia),
  4. traumatic
  5. All others who have an anatomic or known biochemical lesion.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with idiopathic seizure disorders under age 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-02 (Actual); Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chetanbabu M Patel, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospitals and Clinics, Kansas City, Missouri, United States

REFERENCES:
- [Background] Hsu BY, Kelly A, Thornton PS, Greenberg CR, Dilling LA, Stanley CA. Protein-sensitive and fasting hypoglycemia in children with the hyperinsulinism/hyperammonemia syndrome. J Pediatr. 2001 Mar;138(3):383-9. doi: 10.1067/mpd.2001.111818. PMID 11241047
- [Background] Hauser WA. The prevalence and incidence of convulsive disorders in children. Epilepsia. 1994;35 Suppl 2:S1-6. doi: 10.1111/j.1528-1157.1994.tb05932.x. PMID 8275976
- [Background] Sperling MA, Menon RK. Differential diagnosis and management of neonatal hypoglycemia. Pediatr Clin North Am. 2004 Jun;51(3):703-23, x. doi: 10.1016/j.pcl.2004.01.014. PMID 15157593
- [Background] Vilke GM, Castillo EM, Ray LU, Murrin PA, Chan TC. Evaluation of pediatric glucose monitoring and hypoglycemic therapy in the field. Pediatr Emerg Care. 2005 Jan;21(1):1-5. doi: 10.1097/01.pec.0000150980.94571.10. PMID 15643315
- [Background] Valencia I, Sklar E, Blanco F, Lipsky C, Pradell L, Joffe M, Legido A. The role of routine serum laboratory tests in children presenting to the emergency department with unprovoked seizures. Clin Pediatr (Phila). 2003 Jul-Aug;42(6):511-7. doi: 10.1177/000992280304200605. PMID 12921452
- [Background] Hirtz D, Ashwal S, Berg A, Bettis D, Camfield C, Camfield P, Crumrine P, Elterman R, Schneider S, Shinnar S. Practice parameter: evaluating a first nonfebrile seizure in children: report of the quality standards subcommittee of the American Academy of Neurology, The Child Neurology Society, and The American Epilepsy Society. Neurology. 2000 Sep 12;55(5):616-23. doi: 10.1212/wnl.55.5.616. PMID 10980722
- [Background] Raizen DM, Brooks-Kayal A, Steinkrauss L, Tennekoon GI, Stanley CA, Kelly A. Central nervous system hyperexcitability associated with glutamate dehydrogenase gain of function mutations. J Pediatr. 2005 Mar;146(3):388-94. doi: 10.1016/j.jpeds.2004.10.040. PMID 15756227
- [Background] Hauser WA. Seizure disorders: the changes with age. Epilepsia. 1992;33 Suppl 4:S6-14. doi: 10.1111/j.1528-1157.1992.tb06222.x. PMID 1425495
- [Background] Melegh B, Pap M, Morava E, Molnar D, Dani M, Kurucz J. Carnitine-dependent changes of metabolic fuel consumption during long-term treatment with valproic acid. J Pediatr. 1994 Aug;125(2):317-21. doi: 10.1016/s0022-3476(94)70218-7. PMID 8040784
- [Background] Nishida N, Sugimoto T, Araki A, Woo M, Sakane Y, Kobayashi Y. Carnitine metabolism in valproate-treated rats: the effect of L-carnitine supplementation. Pediatr Res. 1987 Nov;22(5):500-3. doi: 10.1203/00006450-198711000-00003. PMID 3120144
- [Background] al-Hosani H, Salah M, Saade D, Osman H, al-Zahid J. United Arab Emirates National Newborn Screening Programme: an evaluation 1998-2000. East Mediterr Health J. 2003 May;9(3):324-32. PMID 15751925
- [Background] Schweitzer-Krantz S. Early diagnosis of inherited metabolic disorders towards improving outcome: the controversial issue of galactosaemia. Eur J Pediatr. 2003 Dec;162 Suppl 1:S50-3. doi: 10.1007/s00431-003-1352-2. Epub 2003 Nov 12. PMID 14614623